CLINICAL TRIAL: NCT05030155
Title: Evaluation of MEpolizumab-based Regimen Compared to Conventional Therapeutic Strategy For Remission Induction In Patients With Eosinophilic Granulomatosis With Polyangiitis. Prospective, Randomized, Controlled, Double-blind Study
Brief Title: Study of Mepolizumab-based Regimen Compared to Conventional Therapeutic Strategy in Patients With Eosinophilic Granulomatosis With Polyangiitis (E-merge)
Acronym: E-merge
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Vasculitis Study Group (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D20180135; 2020-003318-10 (EudraCT Number)
Record Dates: First submitted 2021-07-31; First posted 2021-09-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis
Keywords: Eosinophilic Granulomatosis with Polyangiitis; Mepolizumab; Remission induction; Conventional therapeutic
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — mepolizumab; Cyclophosphamide; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with FFS=0 - Mepolizumab (Experimental): Mepolizumab 300mg every 4 weeks until D336
  Interventions: Drug: Mepolizumab
- Patients with FFS=0 - Placebo (Placebo Comparator): Placebo of Mepolizumab every 4 weeks until D336
  Interventions: Drug: Placebo
- Patients with FFS≥1 - Mepolizumab (Experimental): Mepolizumab 300mg every 4 weeks until D336 and placebo of Azathioprine 1mg/kg/day from D126 until D360 and placebo of cyclophosphamide/mesna at D1, D15, D28, D56, D84 and D112
  Interventions: Drug: Mepolizumab; Drug: Placebo
- Patients with FFS≥1 - Placebo (Placebo Comparator): Placebo of Mepolizumab every 4 weeks until D336, cyclophosphamide and mesna at D1, D15, D28, D56, D84 and D112 and Azathioprine 1mg/kg/day from D126 until D360
  Interventions: Drug: cyclophosphamide/azathioprine; Drug: Placebo

INTERVENTIONS:
Drug: Mepolizumab — 300 mg/month subcutaneous
  Arms: Patients with FFS=0 - Mepolizumab; Patients with FFS≥1 - Mepolizumab
Drug: cyclophosphamide/azathioprine — Patients with FFS≥1 will receive cyclophosphamide then azathioprine
  Arms: Patients with FFS≥1 - Placebo
Drug: Placebo — Patients with FFS=0 will receive placebo
  Arms: Patients with FFS=0 - Placebo; Patients with FFS≥1 - Mepolizumab; Patients with FFS≥1 - Placebo

SUMMARY:
The purpose of this study is to compare mepolizumab-based regimen to conventional therapeutic strategy for remission induction in patients with Eosinophilic Granulomatosis with Polyangiitis.

DETAILED DESCRIPTION:
Eosinophilic granulomatosis with polyangiitis (EGPA), formerly called Churg-Strauss syndrome, is a rare systemic small-vessel vasculitis, associated with asthma and blood and tissue eosinophilia. EGPA belongs to the group of antineutrophil cytoplasmic antibody (ANCA)-associated vasculitides (AAV), and commonly involves upper and lower respiratory tracts, the lungs, the peripheral nerve and the heart.

Therapeutic management is based on glucocorticoids alone or in combination with conventional immunosuppressive agents, mainly azathioprine, methotrexate or cyclophosphamide, according to disease severity assessed by the Five Factor Score.

Such treatments, in addition to their common side effects, are frequently insufficiently effective to control chronic asthma and/or rhinosinusitis, requiring long-term high-dose corticosteroids. Because EGPA shares common pathophysiological features with eosinophilic disorders and asthma, new therapeutic options used in these conditions could be of interest, in particular mepolizumab, a monoclonal anti-interleukin (IL)-5 antibody, which has shown promising results in two small preliminary studies to control disease activity and decrease glucocorticoids in cortico-dependant patients. In addition, mepolizumab has been recently evaluated in a prospective trial, the MIRRA trial, targeting a small niche of patients, i.e. those with corticodependent asthma unable to achieve disease control with low dose of glucocorticoids. Results published revealed that mepolizumab led to significantly more accrued weeks of remission than placebo (28% vs. 3% of the participants had ≥24 weeks of accrued remission; odds ratio, 5.91; 95% confidence interval [CI], 2.68 to 13.03; P<0.001) and a higher percentage of participants in remission at both week 36 and week 48 (32% vs. 3%; odds ratio, 16.74; 95% CI, 3.61 to 77.56; P<0.001).

However, these studies did not evaluate the interest of mepolizumab during EGPA flare associating asthma, eosinophilic and vasculitis lesions, in order to induce remission of the disease and rapidly decrease and discontinue glucocorticoids.

Also, recent pathophysiological date strongly support in addition to previous therapeutic studies the major interest to target IL-5 as soon as EGPA is diagnosed: 1) genetic association studies demonstrated that polymorphisms in the IL-5 pathway are associated with EGPA in comparison with controls, 2) increased expression of IL-5 in mice model are able to induce vasculitis lesions as observed in the human diseases.

Patients will receive a standardized glucocorticoid tapering schedule. From day 28 post-baseline onwards, if the subject's BVAS=0 their oral prednisone dose should be tapered downwards. A standardized glucocorticoid tapering schedule provided in the protocol enables a reduction in oral prednisone dose every 2 weeks, with the intention of achieving a prednisone dose of 4 mg/day or less. Once a subject has achieved a dose of 4 mg/day prednisone, the investigator is encouraged to continue tapering downwards, if clinically warranted, at dose increments of 1.0 mg every week.

Upwards dose adjustments within the 0-4.0 mg range are permitted without necessarily being considered a relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of EGPA independently of ANCA status,
* Patients aged of 18 years or older,
* Patients with newly-diagnosed disease or relapsing disease at the time of screening, with an active disease defined as a Birmingham Vasculitis Activity Score (BVAS) ≥3,
* Patients within the first 21 days following initiation/increase of corticosteroids at a dose ≤ 1 mg/kg/day (pulses of methylprednisolone before oral corticosteroid therapy are authorized)
* Patients having given their written informed consent prior to participation in the study.
* Patients affiliated with social security or CMU (profit or being entitled)

Exclusion Criteria:

* Patients with GPA, MPA, or other vasculitis, defined by the ACR criteria and/or the Chapel Hill Consensus Conference,
* Patients with vasculitis in remission of the disease defined as a BVAS <3
* Patients with severe cardiac failure defined as class IV in New York Heart Association
* Patients with acute infections or chronic active infections (including HIV, HBV or HCV and checked in the last 12 months),
* Patients with active cancer or recent cancer (<5 years), except basocellular carcinoma and prostatic cancer of low activity controlled by hormonal treatment,
* Pregnant women and lactation. Patients with childbearing potential should have reliable contraception for the 12 months duration of the study,
* Patients with EGPA who have already been treated with mepolizumab within the previous 12 months,
* Patients with hypersensitivity to a monoclonal antibody or biologic agent,
* Patients with contraindication to use mepolizumab, cyclophosphamide, mesna, azathioprine or maintenance therapy used for vasculitis,
* Patients with other uncontrolled diseases, including drug or alcohol abuse, severe psychiatric diseases, that could interfere with participation in the trial according to the protocol,
* Patients included in other investigational therapeutic study within the previous 3 months,
* Patients suspected not to be observant to the proposed treatments,
* Patients who have white blood cell count ≤4,000/mm3,
* Patients who have platelet count ≤100,000/mm3,
* Patients who have ALT or AST level greater that 3 times the upper limit of normal that cannot be attributed to underlying EGPA disease,
* Patients unable to give written informed consent prior to participation in the study
* Patients under tutorship or curatorship and protected adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who achieved a prednisone dose of 4.0 mg or less per day at day 168, without experiencing a relapse | Day 168
  EGPA relapse will be defined as worsening or persistence of active disease since the last visit characterized by: a) active vasculitis (BVAS >0); OR b) active asthma symptoms; OR c) active nasal and/or sinus disease, warranting: i) an increased dose of prednisone compared to previous dosage and at least >4 mg/day prednisone total daily dose or equivalent; OR ii) an increased dose or addition of immunosuppressive therapy; OR iii) hospitalisation related to EGPA worsening. A BVAS evaluation will be conducted at the time of a relapse, or as soon as possible afterwards

SECONDARY OUTCOMES:
Prednisone dosage at days 168 and 364 | Days 168 and 364
Area under the curve for corticosteroids at days 168 and 364 | Days 168 and 364
Proportion of participants with a prednisone dose of 4.0 mg or less per day for 0 weeks | Days 168 and 364
Proportion of participants with a prednisone dose of 4.0 mg or less per day for more than 0 weeks but less than 4 weeks | Days 168 and 364
Proportion of participants with a prednisone dose of 4.0 mg or less per day for more than 4 weeks but less than 12 weeks | Days 168 and 364
Proportion of participants with a prednisone dose of 4.0 mg or less per day for at least 12 weeks | Days 168 and 364
Proportion of participants with a prednisone dose of 4.0 mg or less per day at both days 168 and 364. | Day 364
Proportion of participants experiencing a relapse | Day 364
  EGPA relapse will be defined as worsening or persistence of active disease since the last visit characterized by: a) active vasculitis (BVAS >0); OR b) active asthma symptoms; OR c) active nasal and/or sinus disease, warranting: i) an increased dose of prednisone compared to previous dosage and at least >4 mg/day prednisone total daily dose or equivalent; OR ii) an increased dose or addition of immunosuppressive therapy; OR iii) hospitalisation related to EGPA worsening. A BVAS evaluation will be conducted at the time of a relapse, or as soon as possible afterwards
Number of relapse during the study period | Day 364
  EGPA relapse will be defined as worsening or persistence of active disease since the last visit characterized by: a) active vasculitis (BVAS >0); OR b) active asthma symptoms; OR c) active nasal and/or sinus disease, warranting: i) an increased dose of prednisone compared to previous dosage and at least >4 mg/day prednisone total daily dose or equivalent; OR ii) an increased dose or addition of immunosuppressive therapy; OR iii) hospitalisation related to EGPA worsening. A BVAS evaluation will be conducted at the time of a relapse, or as soon as possible afterwards.
Time from inclusion to first relapse | Day 364
Number of adverse events that result in the cessation of further injections | Day 364
  Number of adverse events is expressed as adverse events according to the CTCAE toxicity grading system per patient-year at days 168 and 364 for the following adverse events combined: death (all causes), grade 2 or higher leukopenia or thrombocytopenia, grade 3 or higher infections, hemorraghic cystitis, malignancies, venous thromboembolic events, hospitalization resulting either from the disease or from a complication due to the study treatment, injection reactions (within 24 hours of injection).
Vasculitis Damage Index (VDI) | Days 168 and 364
HAQ questionnaire | Days 168 and 364
SF-36 questionnaire | Days 168 and 364
Evolution of ANCA titers (in UI/mL) and correlation with clinical events during follow-up | Day 364
Evolution of eosinophils (in x10^9/L) and correlation with clinical events during follow-up | Day 364

CONTACTS AND LOCATIONS:
Overall Officials: Loic GUILLEVIN, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Interne, Centre de référence " Maladies systémiques et autoimmunes rares, en particulier Vascularites nécrosantes et Sclérodermies systémiques "Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No